CLINICAL TRIAL: NCT05371496
Title: Evaluation of the Cardiac and Metabolic Effects of Semaglutide in Heart Failure With Preserved Ejection Fraction (CAMEO-SEMA) A Phase II, Prospective, Double-Blind Randomized Trial
Brief Title: Cardiac and Metabolic Effects of Semaglutide in Heart Failure With Preserved Ejection Fraction
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Barry Borlaug, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-000522
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Cardiomyopathy; Heart Failure With Preserved Ejection Fraction (HFpEF); Obesity
MeSH Terms: conditions — Cardiomyopathies; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide Treatment (Active Comparator): Subjects will receive Semaglutide once weekly in addition to counselling on healthy lifestyle intervention
  Interventions: Drug: Semaglutide; Behavioral: Counselling on healthy lifestyle intervention
- Placebo Treatment (Placebo Comparator): Subjects will receive matching placebo once weekly in addition to counselling on healthy lifestyle intervention
  Interventions: Drug: Placebo; Behavioral: Counselling on healthy lifestyle intervention

INTERVENTIONS:
Drug: Semaglutide — 3.0 mg/ml (titrated to 2.4 mg) subcutaneous once weekly for 12 months
  Arms: Semaglutide Treatment
Drug: Placebo — Matched placebo with no active drug once weekly for 12 months
  Arms: Placebo Treatment
Behavioral: Counselling on healthy lifestyle intervention — All participants will receive counselling on healthy lifestyle intervention including limiting consumption of salt, red meat, saturated or trans fats, sweets, and sugar-sweetened beverages, and how to restrict calorie intake (500 kcal/day deficit) in consultation with a trained study dietician. Regular physical activity >150 minutes per week will be encouraged.

SUMMARY:
The purpose of this research is to find out if an aggressive intervention to lose weight, will improve symptoms in patients with obesity-related cardiomyopathy, which is also known as the obese phenotype of heart failure with preserved ejection fraction (HFpEF).

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30.0 kg/m2.
* NYHA Class II-IV.
* LVEF ≥ 50 % within the preceding year.
* No hospitalizations due to heart failure in the preceding 30 days.
* At least one of the following:

  1. Mean PCWP ≥ 15 mmHg or left ventricular end diastolic pressure (LVEDP) ≥ 15 mmHg documented during catheterization at rest, or PCWP or LVEDP ≥ 25 mmHg documented during catheterization at exercise.
  2. If BMI < 35.0: NT-proBNP ≥ 220 pg/mL (for patients with sinus rhythm) or NT-proBNP ≥ 660 pg/mL (for patients with persistent/permanent atrial fibrillation); if BMI ≥ 35.0: NT-proBNP ≥ 125 pg/mL (for patients in sinus rhythm) or NT-proBNP ≥ 375 pg/mL (for patients with persistent/ permanent atrial fibrillation) at screening (NT-proBNP analyzed by the central laboratory) in combination with at least one of the following (documented by echocardiography within 12 months prior to or at screening): i. Septal é < 7 cm/sec or lateral é < 10 cm/sec or average E/é ≥ 15. ii. PA systolic pressure > 35 mmHg. iii. Left atrial (LA) enlargement (LA width ≥ 3.8 cm or LA length ≥ 5.0 cm or LA area ≥ 20.0 cm2 or LA volume ≥ 55 mL or LA volume index ≥ 29 mL/m2). iv. LV hypertrophy with septal thickness or posterior wall thickness ≥ 1.2 cm
  3. Hospitalization with a primary diagnosis of decompensated heart failure which required intravenous (IV) loop diuretic treatment, within the previous 12 months in combination with at least two of the following (documented by echocardiography within 12 months prior to or at screening): i. Septal é < 7 cm/sec or lateral é < 10 cm/sec or average E/é ≥ 15. ii. PA systolic pressure > 35 mmHg. iii. LA enlargement (LA width ≥ 3.8 cm or LA length ≥ 5.0 cm or LA area ≥ 20.0 cm2 or LA volume ≥ 55 mL or LA volume index ≥ 29 mL/m2). iv. LV hypertrophy with septal thickness or posterior wall thickness ≥ 1.2 cm. v. Ongoing use of diuretic therapy for at least 30 days prior to screening.

Exclusion Criteria:

Cardiovascular-related:

* Myocardial infarction, stroke, hospitalization for heart failure, unstable angina pectoris or transient ischemic attack within 30 days prior to the day of screening.
* Systolic blood pressure > 160 mmHg at screening.
* Planned coronary, carotid or peripheral artery revascularization.
* Any other condition judged by the investigator to be the primary cause of dyspnea (such as heart failure due to restrictive cardiomyopathy or infiltrative conditions (e.g., amyloidosis), hypertrophic obstructive cardiomyopathy, primary pulmonary arterial hypertension, chronic obstructive pulmonary disease, right heart failure due to pulmonary disease, complex congenital heart disease, anemia, or more than moderate mitral or aortic heart valve disease).

  * Amyloid cardiomyopathy may be present in 5-15% of patients presenting with the clinical syndrome of HFpEF,60-62 and patients with amyloid may respond differently to WL intervention. To enhance the scientific rigor of the trial by ensuring a homogenous population of true primary HFpEF, we will carefully evaluate for the presence of amyloid using the approach outlined in a recent scientific statement from the AHA,63 which is also consistent with our current clinical practice.
  * Specifically, potential participants will be evaluated for clues or risk factors for underlying cardiac amyloid including intolerance to antihypertensives, hypotension, orthostatic intolerance, persistent low-grade elevation in troponin, low QRS voltage on ECG, unexplained AV block or prior pacemaker, unexplained LV or RV wall thickening, impaired LV global longitudinal strain with apical sparing by echocardiography, family history of cardiomyopathy, neuropathy, autonomic dysfunction, carpal tunnel syndrome, lumbar spinal stenosis, family history of polyneuropathy, or black race. Patients with these risk factors will undergo screening evaluation for amyloid prior to consent in CAMEO-SEMA as part of best clinical practice. This includes screening for monoclonal light chain as first step, followed by hematology consultation if the screen is positive. Patients with risk factors but no monoclonal light chain will then undergo Tc-99m-PYP scan to rule out cardiac amyloid.

Obesity-related:

* Bariatric surgery prior to screening within 5 years of screening or planned bariatric surgery within the trial time course.
* A self-reported change in body weight > 5 kg (11 lbs) within 90 days before screening irrespective of medical records.

Glycemia-related:

* HbA1c ≥ 10.0% based on latest available value from medical records, not older than 3 months
* History of type 1 diabetes (history of gestational diabetes is allowed).
* Treatment with any GLP-1 receptor agonist within 90 days prior to the day of screening.

General health and safety:

* Personal or first-degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma.
* Presence of acute pancreatitis within the last 180 days prior to screening.
* History or presence of chronic pancreatitis.
* End-stage renal disease or chronic or intermittent hemodialysis or peritoneal dialysis.
* Presence or history of malignant neoplasm within 5 years prior to the day of screening. Basal and squamous cell cancer and any carcinoma in-situ are allowed.
* Known or suspected hypersensitivity to trial product(s) or related products.
* Participation in any clinical trial of an approved or non-approved device for the treatment of heart failure or obesity within 30 days before screening.
* Receipt of any investigational medicinal product within 30 days before screening.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method.
* Major surgery scheduled for the duration of the trial, affecting walking ability in the opinion of the investigator.
* Any disorder, including severe psychiatric disorder, suicidal behavior within 90 days before screening, and suspected drug abuse, which in the investigator´s opinion might jeopardize subject´s safety or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Capillary Wedge Pressure (PCWP) | Baseline, 12 months
  Change in PCWP during exercise, reported in mmHG

SECONDARY OUTCOMES:
Trans-cardiac uptake of free fatty acids (FFA) at rest | Baseline, 12 months
  Change in trans-cardiac uptake of FFA will be measured using arterial and coronary sinus blood samples collected at rest during cardiac catheterization procedure.
Trans-cardiac uptake of free fatty acids (FFA) during exercise | Baseline, 12 months
  Change in trans-cardiac uptake of FFA will be measured using arterial and coronary sinus blood samples collected during the exercise portion of the cardiac catheterization procedure.
Trans-cardiac uptake of glucose at rest | Baseline, 12 months
  Change in trans-cardiac uptake of glucose will be measured using arterial and coronary sinus blood samples collected at rest during the cardiac catheterization procedure.
Trans-cardiac uptake of glucose during exercise | Baseline, 12 months
  Change in trans-cardiac uptake of glucose will be measured using arterial and coronary sinus blood samples collected during the exercise portion of the cardiac catheterization procedure.
Trans-cardiac uptake of ketone bodies at rest | Baseline, 12 months
  Change in trans-cardiac uptake of ketone bodies will be measured using arterial and coronary sinus blood samples collected at rest during the cardiac catheterization procedure.
Trans-cardiac uptake of ketone bodies during exercise | Baseline, 12 months
  Change in trans-cardiac uptake of ketone bodies will be measured using arterial and coronary sinus blood samples collected during the exercise portion of the cardiac catheterization procedure.
Left ventricular (LV) global longitudinal strain | Baseline, 12 months
  Change in LV global longitudinal strain will be assessed by echocardiography conducted during the cardiac catheterization procedure
Left Atrial (LA) reservoir strain | Baseline, 12 months
  Change in LA reservoir strain will be assessed by echocardiography conducted during the cardiac catheterization procedure
Right Ventricular (RV) free wall strain | Baseline, 12 months
  Change in RV free wall strain will be assessed by echocardiography conducted during the cardiac catheterization procedure
Myocardial mass | Baseline, 12 months
  Change in myocardial mass will be measured by CMR imaging.
Myocardial volume | Baseline, 12 months
  Change in myocardial volume will be measured by CMR imaging.
Myocardial fat content | Baseline, 12 months
  Change in myocardial fat content will be measured by CMR imaging.
Body fat mass | Baseline, 12 months
  Change in body fat mass will be measured using dual X-ray absorptiometry (DEXA)
Visceral fat content | Baseline, 12 months
  Change in visceral fat content will be measured using limited abdominal MRI
Total blood volume | Baseline, 12 months
  Change in total blood volume will be assessed by using the radiolabeled iodinated albumin (131I, 5-25 μCu) indicator dilution technique (BVA-100 Blood Volume Analyzer, Daxor Corp, NY).
Total plasma volume | Baseline, 12 months
  Change in total plasma volume will be assessed by using the radiolabeled iodinated albumin (131I, 5-25 μCu) indicator dilution technique (BVA-100 Blood Volume Analyzer, Daxor Corp, NY).
Change in Quality of Life (QOL) as assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline, 12 months
  KCCQ was a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 (worst) and 100 (the best possible status), where the higher score reflected better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No